CLINICAL TRIAL: NCT06452719
Title: Letrozole and Misoprostol for Early Pregnancy Loss Management: A Prospective Pilot Cohort Study
Brief Title: Letrozole and Misoprostol for Early Pregnancy Loss Management
Acronym: LeMi
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 855835
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Early Pregnancy Loss; Miscarriage in First Trimester; Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Letrozole; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Letrozole & Misprostol (Experimental): Letrozole 10 mg orally daily for three consecutive days followed by misoprostol 800 mcg vaginally within 24 hours of final letrozole dose
  Interventions: Drug: Letrozole; Drug: Misoprostol

INTERVENTIONS:
Drug: Letrozole — Letrozole 10 mg orally daily for three consecutive days
Drug: Misoprostol — Misoprostol 800 mcg vaginally within 24 hours of final letrozole dose

SUMMARY:
A pilot cohort study to preliminarily investigate the efficacy of pretreatment with letrozole 10 mg daily for three consecutive days followed by treatment with misoprostol 800 mcg vaginally for medical management of early pregnancy loss in a US population. Patients will be followed to assess efficacy of this treatment regimen, as well as additional interventions needed, side effects, adverse events, and patient acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in the informed consent process and provide a signed and dated consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Access to working mobile phone
* English-speaking
* Age 18 years or older
* Confirmed diagnosis of intrauterine embryonic/fetal demise or anembryonic gestation (ultrasound examination demonstrates a fetal pole without cardiac activity measuring between 5.3 and 40 mm or an abnormal growth pattern diagnostic of early pregnancy failure)

Exclusion Criteria:

* Incomplete or inevitable abortion
* Contraindication of allergy to letrozole or misoprostol
* Unable to return for clinic-based follow-up
* Twin or multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy | Visit 2 (Days 10-11)
  Absence of gestational sac on transvaginal ultraound

SECONDARY OUTCOMES:
Acceptability | 30 days
  Participant assessment of treatment (Positive / Neutral / Negative), Likelihood to recommend this method of treatment to a friend (Yes / No)

CONTACTS AND LOCATIONS:
Locations (1):
- PEACE / Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No